CLINICAL TRIAL: NCT00605566
Title: Tailored-dose Sorafenib Plus Metronomic Cyclophosphamide in Advanced Neuroendocrine Tumors (NET): a Phase II Clinical Trial Based on Individual Pharmacodynamic Assessment
Brief Title: Efficacy Study of Sorafenib and Cyclophosphamide to Treat Neuroendocrine Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SOR-NET-001
Record Dates: First submitted 2008-01-18; First posted 2008-01-31 (Estimated); Results first posted 2019-02-19 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2018-10

CONDITIONS: Neuroendocrine Tumors
Keywords: Neuroendocrine; sorafenib; cyclophosphamide; pharmacodynamic
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Sorafenib; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- I (Experimental): Patients will receive sorafenib and cyclophosphamide.
  Interventions: Drug: Sorafenib; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Sorafenib — During a run-in period, patient will start taking 50 mg QD of oral cyclophosphamide and 200 mg BID of sorafenib. On day 8 of run-in the patient will be evaluated for toxicity. In the absence of toxicity, the patient will be escalated to sorafenib 400 mg BID and continue on daily 50 mg of cyclophosphamide, or the patient will be informed to continue on sorafenib 200 mg BID and cyclophosphamide 50 mg QD. Dose escalation procedure will be repeated every 2 weeks until unable to tolerate the study drug, or a maximum of 800 mg BID is reached, or achievement of > 90% inhibition of phosphorylation of PDGFR/Raf axis in PBMC. After "run-in" period, patient begins cycle 1, each cycle will last 28 days. Both cyclophosphamide and sorafenib will be taken orally.
  Other Names: BAY 43-9006
Drug: Cyclophosphamide — During a run-in period, patient will start taking 50 mg QD of oral cyclophosphamide and 200 mg BID of sorafenib. On day 8 of run-in the patient will be evaluated for toxicity. In the absence of toxicity, the patient will be escalated to sorafenib 400 mg BID and continue on daily 50 mg of cyclophosphamide, or the patient will be informed to continue on sorafenib 200 mg BID and cyclophosphamide 50 mg QD. Dose escalation procedure will be repeated every 2 weeks until unable to tolerate the study drug, or a maximum of 800 mg BID is reached, or achievement of > 90% inhibition of phosphorylation of PDGFR/Raf axis in PBMC. After "run-in" period, patient begins cycle 1, each cycle will last 28 days. Both cyclophosphamide and sorafenib will be taken orally.
  Other Names: Cytoxan

SUMMARY:
This is a phase II clinical trial to assess the efficacy of the combination of metronomic cyclophosphamide and tailored sorafenib dosing in advanced, progressive NET. NET are highly vascular tumors, and high VEGF expression has been correlated with worse clinical and pathological characteristics as well as poor prognosis. A novel antiangiogenic approach relies on targeting not only the endothelial cells but also rendering them more sensitive to VEGFR blockade by achieving pericyte detachment. In this study, the dose of sorafenib will be titrated up to a maximum of 800mg BID based on patients' toxicity and on a novel pharmacodynamic assay that measures inhibition of molecular target(PDGFR) in patients' peripheral blood mononuclear cells. Dual VEGFR targeting is achieved by administering sorafenib plus metronomic low dose cyclophosphamide.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed neuroendocrine tumors
* Progressive and measurable metastatic disease
* Patients must not have disease that is currently amenable to surgery
* Life expectancy of greater than 3 months
* ECOG performance status ≤2
* Patients must have normal organ and marrow function
* Negative pregnancy test; agreement to use adequate birth control

Exclusion Criteria:

* Patients receiving chemotherapy or radiotherapy within last 4 weeks
* Patients that had received Sorafenib for advanced NET(neuroendocrine tumors) are not allowed
* Any other investigational agents within 4 weeks of study
* Patients with known brain metastases
* History of allergic reactions to compounds of similar chemical/biologic composition to sorafenib or cyclophosphamide
* Concurrent cancer from another primary site requiring treatment within the past 3 years
* Uncontrolled intercurrent illness
* Pregnant women and women who are breastfeeding
* HIV-positive patients receiving combination anti-retroviral therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-01; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lillian Siu, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from January 2008 to October 2010.
Groups:
- Sorafenib and Cyclophosphamide: Patients will receive sorafenib and cyclophosphamide.
  sorafenib and cyclophosphamide: During a run-in period, patient will start taking 50 mg QD of oral cyclophosphamide and 200 mg BID of sorafenib. On day 8 of run-in the patient will be evaluated for toxicity. In the absence of toxicity, the patient will be escalated to sorafenib 400 mg BID and continue on daily 50 mg of cyclophosphamide, or the patient will be informed to continue on sorafenib 200 mg BID and cyclophosphamide 50 mg QD. Dose escalation procedure will be repeated every 2 weeks until unable to tolerate the study drug, or a maximum of 800 mg BID is reached, or achievement of > 90% inhibition of phosphorylation of PDGFR/Raf axis in PBMC. After "run-in" period, patient begins cycle 1, each cycle will last 28 days. Both cyclophosphamide and sorafenib will be taken orally.
Period: Overall Study
Arm/Group | Sorafenib and Cyclophosphamide
Started | 22
Completed | 19
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Clinical deterioration | 1
Not completed — Poor compliance in run-in period | 1

BASELINE CHARACTERISTICS:
Groups:
- Sorafenib Plus Cyclophosphamide: Patients will receive sorafenib and cyclophosphamide.
  sorafenib and cyclophosphamide: During a run-in period, patient will start taking 50 mg QD of oral cyclophosphamide and 200 mg BID of sorafenib. On day 8 of run-in the patient will be evaluated for toxicity. In the absence of toxicity, the patient will be escalated to sorafenib 400 mg BID and continue on daily 50 mg of cyclophosphamide, or the patient will be informed to continue on sorafenib 200 mg BID and cyclophosphamide 50 mg QD. Dose escalation procedure will be repeated every 2 weeks until unable to tolerate the study drug, or a maximum of 800 mg BID is reached, or achievement of > 90% inhibition of phosphorylation of PDGFR/Raf axis in PBMC. After "run-in" period, patient begins cycle 1, each cycle will last 28 days. Both cyclophosphamide and sorafenib will be taken orally.
Arm/Group | Sorafenib Plus Cyclophosphamide
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 5
Age, Continuous [Median (Full Range); unit: years] | 58 [32 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 12

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Combination Sorafenib Plus Metronomic Cyclophosphamide in Advanced, Progressive NET, as Measured by the Objective Response Rate (ORR).
Description: Objective response (complete and partial) evaluated using RECIST criteria. Complete response (CR): disappearance of all clinical and radiological evidence of tumour (both target and non-target).
  Partial response (PR): at least a 30% decrease in the sum of longest diameter of target lesions.
Time Frame: Assessed from start of study treatment until death or disease progression, whichever occurs first up to 7 years
Population: 19 out of 22 patients were evaluable for response.
Measure: Count of Participants; unit: Participants
Arm/Group | Sorafenib and Cyclophosphamide
Number analyzed (Participants) | 19
Participants | 1

2. Primary Outcome: Association Between p-Shift Changes and Treatment Efficacy of Individual Dose Adjustment of Sorafenib
Description: A phosphoshift (pShift) flow cytometry-based test that measures RAF signal transduction capacity in peripheral blood cells was used in order to predict clinical course and/or guide individual dose-titration. Positive pShift values denote stimulation of RAF signal transduction, whereas negative pShift values denote inhibition of RAF signal transduction as measured by flow-cytometry.
  Associations between pShift changes and treatment efficacy were measured using progression-free survival (PFS) and overall survival (OS).
Time Frame: Assessed from start of study treatment until death, assessed up to 7 years.
Population: 6 patients experienced a pharmacodynamic pShift change that was classified as positive, 16 experienced a negative pShift.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sorafenib and Cyclophosphamide
Number analyzed (Participants) | 22
months
  PFS in patients with a negative pShift result: number analyzed (Participants) | 16
  PFS in patients with a negative pShift result | 2.8 [1.8 to 6.7]
  PFS in patients with a positive pShift result: number analyzed (Participants) | 6
  PFS in patients with a positive pShift result | 14.9 [3 to NA] — Not reached
  OS for patients with a negative pShift: number analyzed (Participants) | 16
  OS for patients with a negative pShift | 6.4 [2.8 to 6.4]
  OS for patients with a positive pShift: number analyzed (Participants) | 6
  OS for patients with a positive pShift | 21.3 [7.9 to NA] — Not reached

3. Secondary Outcome: Progression-free Survival (PFS)
Description: Progressive disease (PD): at least a 20% increase in the sum of the longest diameter of measured lesions.
Time Frame: Assessed from start of study treatment until death or disease progression, whichever occurs first up to 7 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sorafenib and Cyclophosphamide
Number analyzed (Participants) | 22
months | 3 [2 to 10.7]

4. Secondary Outcome: Overall Survival (OS)
Time Frame: Assessed from start of study treatment until death, assessed up to 7 years.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sorafenib and Cyclophosphamide
Number analyzed (Participants) | 22
months | 11.7 [4.3 to NA] — Not reached

5. Secondary Outcome: 1-year Survival Rate
Description: Survival rate at 1 year.
Time Frame: 1 year
Measure: Number; unit: percentage of participants
Arm/Group | Sorafenib and Cyclophosphamide
Number analyzed (Participants) | 22
percentage of participants | 45

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over a total of 160 treatment cycles (1 cycle = 28 days) for all study participants, for as long as 7 years.
Arm/Group | Sorafenib Plus Cyclophosphamide
Serious Adverse Events (participants affected / at risk) | 11/22
Other Adverse Events (participants affected / at risk) | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sorafenib Plus Cyclophosphamide (N=22)
Ileal perforation (Gastrointestinal disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 2 (2)
Flushing (Vascular disorders) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Protein Urine Positive (Renal and urinary disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Weight Gain (Investigations) | 1 (1)
Disease progression (General disorders) | 1 (1)
Bilirubin increased (Investigations) | 1 (1)
Lipase increased (Investigations) | 2 (2)
Amylase increased (Investigations) | 1 (1)
Fever (General disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib Plus Cyclophosphamide (N=22)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 10
Dysgeusia (Nervous system disorders) | 5
Hypertension (Vascular disorders) | 3
Fatigue (General disorders) | 9
Diarrhoea (Gastrointestinal disorders) | 12
Alopecia (Skin and subcutaneous tissue disorders) | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 11
Rash (Skin and subcutaneous tissue disorders) | 9
Lymphopenia (Investigations) | 7
Weight loss (Investigations) | 6
Aspartate aminotransferase elevation (Investigations) | 6
Nausea (Gastrointestinal disorders) | 8
Thrombocytopenia (Investigations) | 3
Lipase elevation (Investigations) | 6
Peripheral sensory neuropathy (Nervous system disorders) | 1
Amylase elevation (Investigations) | 5
Vomiting (Gastrointestinal disorders) | 5
Alanine aminotransferase elevation (Investigations) | 3
Hypocalcemia (Metabolism and nutrition disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes